CLINICAL TRIAL: NCT05954559
Title: High Relaxivity Contrast Agent for Cardiac MR in the Myocardial Scar Assessment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00396901
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Fibrosis
MeSH Terms: interventions — gadopiclenol

STUDY DESIGN:
Intervention Model Description: non-randomized cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.05 mmol/kg Elucirem (Experimental): a group that receives 0.05 mmol/kg Elucirem
  Interventions: Drug: Elucirem (Gadopiclenol)
- 0.075 mmol/kg Elucirem (Experimental): A group that receives 0.075 mmol/kg Elucirem
  Interventions: Drug: Elucirem (Gadopiclenol)

INTERVENTIONS:
Drug: Elucirem (Gadopiclenol) — Elucirem (Gadopiclenol) is a new macrocyclic gadolinium-based contrast agent (GBCA) with high relaxivity indicated for use in adults and children aged 2 years and older for contrast-enhanced magnetic resonance imaging.

SUMMARY:
Elucirem (Gadopiclenol) is a new macrocyclic gadolinium-based contrast agent (GBCA) with high relaxivity indicated for use in adults and children aged 2 years and older for contrast-enhanced magnetic resonance imaging. The product was approved in 2022 by FDA to be used to detect and visualize lesions with abnormal vascularity in the central nervous system (brain, spine and associated tissues) and the body (head and neck, thorax, abdomen, pelvis, and musculoskeletal system). However, given its at least twofold higher relaxivity than other GBCAs, the performance of Elucirem in cardiac MR (CMR) has yet to be demonstrated.

The hypothesis for the study: Half dose (0.05mmol/kg) Elucirem is not inferior to double dose (0.2 mmol/kg) Dotarem in the myocardial scar assessment.

All participants will be selected from the investigators previous CMR study cohort with double-dose Dotarem T1 mapping and LGE images. Ten participants without scars will be recruited for the Phase I dose evaluation. Five for 0.05 mmol/kg and five for 0.075 mmol/kg. The investigators have identified 15 participants with LGE findings from double-dose Dotarem CMR acquired in the years 2021, 2022, or earlier years. This study was performed in August 2022. The same protocol will be used for single-dose Elucirem.

DETAILED DESCRIPTION:
Elucirem (Gadopiclenol) is a new macrocyclic gadolinium-based contrast agent (GBCA) with high relaxivity indicated for use in adults and children aged 2 years and older for contrast-enhanced magnetic resonance imaging. The product was approved in 2022 by FDA to be used to detect and visualize lesions with abnormal vascularity in the central nervous system (brain, spine, and associated tissues) and the body (head and neck, thorax, abdomen, pelvis, and musculoskeletal system).

Based on the investigators previous experience with 0.2 mmol/kg Dotarem, the optimal post-contrast T1 for LGE was when the remote myocardium (i.e. area without scar) had T1 of around 400ms at 12 mins post-contrast. The investigators hypothesize that with 0.05 mmol/kg Elucirem, post T1 will recover to 400 ms faster than 12 minutes after injection. It will likely be between 6 to 10 minutes post-contrast. A serial of T1 mapping will provide the information for timing. However, if myocardial T1 were not reduced short enough or recovers to 400 ms in less than 5 minutes post-contrast with 0.05 mmol/kg Elucirem, that is a sign of inadequate dose. Same evaluation will be performed for 0.075 mmol/kg Elucirem. The investigators hypothesize that if 0.05 mmol/kg falls short, 0.075 mmol/kg should be adequate. Since a single dose (0.1 mmol/kg) of Dotarem is proved to be adequate for LGE in many literatures, less Elucirem should be used to demonstrate its benefit.

Study Procedure: It is a non-randomized cohort study. Participants with precious double dose Dotarem CMR will be recruited. The study has two phases. Phase I is to evaluate the optimal dose, 0.05 mmol/kg (N=5) or 0.075 mmol/kg (N=5) by assessing a serial of the myocardial T1 mapping in normal volunteers. T1 mapping will be acquired every 2.5 minutes after injection to 25 minutes post-contrast. Based on the results of Phase I, the optimal dose will be used in the Phase II scar assessment in patients with a scar from a previous double-dose Dotarem study.

ELIGIBILITY:
Inclusion Criteria:

* Participants from previous double-dose Doatrem CMR study who are willing to participate and sign the consent will be enrolled in this study. Participants must be ≥21 years old, less than 120kg, not claustrophobic, and eGFR be 60 and more.

Exclusion Criteria:

* Participants under 21 years old will be excluded. Contraindications or limitations to contrast-enhanced MRI such as self-report of kidney disease, including kidney transplant or kidney surgery, eGFR less than 60, Metal fragments in eyes, brain, or spinal cord, Internal electrical devices such as cochlear implant, spinal cord stimulator, pacemaker, or defibrillator, pregnancy, allergic reaction to gadolinium in the past, claustrophobia, and cardiogenic shock or unstable condition that cannot tolerate the MRI scan will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of half dose of Elucirem to double dose Dotarem | 1-2 years
  Half dose (0.05mmol/kg) Elucirem is not inferior to double dose (0.2 mmol/kg) Dotarem in the myocardial scar assessment.

SECONDARY OUTCOMES:
Post-contrast T1 values | 1-2 years
  Post-contrast T1 values will be measured.
late gadolinium enhancement (LGE), | 1-2 years
  late gadolinium enhancement (LGE) will be measured.
Extracellular volume fraction (ECV) | 1-2 years
  Extracellular volume fraction (ECV) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Lima, Professor, Principal Investigator — MD
Locations (2):
- United States (2):
  - Johns Hopkins Center for Advanced Imaging and Research Science, located in the Science + Technology Park at 1812 Ashland Avenue, Baltimore, MD., Baltimore, Maryland
  - Johns Hopkins School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in Gadolinium Contrast. Data shared will not contain any personal health information (PHI). A statement of work and data use agreement are pre-requisites for data sharing.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication. Data will be made accessible up to 24 months with extensions considered as needed.
Access Criteria: Access provided upon request.